CLINICAL TRIAL: NCT00236665
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study of the Efficacy and Safety of Topiramate in the Treatment of Obese Patients With Mild to Moderate Essential Hypertension
Brief Title: A Study of Efficacy and Safety of Topiramate in the Treatment of Obese Patients With Mild to Moderate Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003727
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Obesity; Hypertension
Keywords: Obesity; Essential Hypertension; Mild Hypertension; Moderate Hypertension; High Blood Pressure
MeSH Terms: conditions — Obesity; Hypertension; Essential Hypertension | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to compare the efficacy and safety of daily topiramate (96mg or 192mg) versus placebo in obese patients with mild to moderate high blood pressure.

DETAILED DESCRIPTION:
Topiramate is not approved for the treatment of obesity. The use of topiramate to reduce weight in obese patients may have the adjunctive benefit of reducing blood pressure in subjects with treated or untreated hypertension, on or off background antihypertensive medications. This double-blind, placebo controlled study investigates the long-term efficacy of topiramate for reduction of weight and blood pressure in obese patients with mild-moderate hypertension, and the safety and tolerability of topiramate in this patient population. The study consists of 4 phases: 6 week run-in phase (2 weeks screening and 4 weeks single-blind placebo), 8 week titration phase (topiramate group will have their dose increased from 16mg/day to either 96mg/day or 192mg/day), 52 week maintenance phase (patients will receive fixed dose of either topiramate or placebo) and 6 week follow-up phase. Beginning at enrollment and throughout the study, all subjects participated in a standardized behavioral modification program which provides subjects with lifestyle and self-management strategies for diet, nutrition and physical activity. Effectiveness will be evaluated by multiple measurements such as change in body weight, sitting diastolic blood pressure, sitting systolic blood pressure, Body Mass Index, number and proportion of treatment responders, volume of left ventricle of the heart as measured by echocardiography, and fasting lipid profile. Safety evaluations (incidence and severity of adverse events, vital signs, 12 lead ECG, clinical laboratory results) will be conducted throughout the study. The study hypothesis is that topiramate is effective in reducing blood pressure in obese patients with mild to moderate hypertension and is well tolerated. During the initial 8 weeks, the dose of topiramate or placebo will be gradually increased to the target doses (either 48mg twice daily or 96mg twice daily by mouth) and the doses will be maintained for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate essential hypertension (sitting diastolic blood pressure >= 90 and < 110 and/or sitting systolic blood pressure >= 140 and < 180)
* Diagnosis of obesity (Body Mass Index >= 27 and < 50 and steady body weight)
* Female patients must be postmenopausal for at least 1 year, surgically incapable of childbearing, practicing abstinence, or practicing an acceptable method of contraception (requires negative pregnancy test)

Exclusion Criteria:

* Prior exposure or known contraindication or hypersensitivity to topiramate
* Pregnancy, nursing or subjects who plan to become pregnant during the study
* Diagnosis of severe hypertension
* History or diagnosis of Diabetes Mellitus
* A history of diastolic or systolic hypertension secondary to a known cause
* Significant cardiovascular or liver disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 531 (Actual)
Dates: Start 2001-03; Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
The percent change in body weight and in sitting diastolic blood pressure from baseline/randomization (Week 0) to Week 60.

SECONDARY OUTCOMES:
Percent change in body weight (from enrollment only), absolute change in body weight, Body Mass Index, sitting systolic and diastolic blood pressure from enrollment and baseline to week 60; safety evaluations during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Tonstad S, Tykarski A, Weissgarten J, Ivleva A, Levy B, Kumar A, Fitchet M. Efficacy and safety of topiramate in the treatment of obese subjects with essential hypertension. Am J Cardiol. 2005 Jul 15;96(2):243-51. doi: 10.1016/j.amjcard.2005.03.053. PMID 16018851